CLINICAL TRIAL: NCT03363087
Title: High Density Scar Guided Atrial Fibrillation Mapping (HD SAGA) / High Density Scar Guided Atrial Fibrillation Mapping StablePoint (HD SAGA S)/ High Density Scar Guided Atrial Fibrillation Mapping HD Grid (HD SAGA H)
Brief Title: High Density Scar Guided Atrial Fibrillation Mapping
Acronym: HD-SAGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Boston Scientific Corporation (Industry); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RHM CAR0523
Record Dates: First submitted 2017-07-28; First posted 2017-12-06 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2022-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Scar; Atrial Fibrillation Ablation; Mapping; Persistent Atrial Fibrillation; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Biatrial automated scar mapping in patients undergoing ablation for atrial fibrillation. Confirmation of scar by pacing in all patients. Collection of impedance data during clinical ablation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mapping (Rhythmia) and ablation (IntellaNav MiFi) (Experimental): Automated high density biatrial scar mapping Pacing confirmation of scar Collection of impedance data during clinical ablation
  Interventions: Device: Mapping and ablation
- Mapping (Rhythmia) and ablation (StablePoint) (Experimental): Automated high density biatrial scar mapping Pacing confirmation of scar Collection of impedance data during clinical ablation Contact force measurements
  Interventions: Device: Mapping and ablation
- Mapping (Precision) (Experimental): Automated high density left atrial mapping in AF and SR in different bipole orientations
  Interventions: Device: Mapping

INTERVENTIONS:
Device: Mapping and ablation — Ultra high density scar mapping Collection of impedance data during ablation
  Arms: Mapping (Rhythmia) and ablation (IntellaNav MiFi); Mapping (Rhythmia) and ablation (StablePoint)
Device: Mapping — Omnipolar mapping of left atrial scar and pulmonary vein isolation lines
  Arms: Mapping (Precision)

SUMMARY:
HD SAGA:

There is increasing evidence that having AF is associated with some scarring of the upper chamber of the heart, the left atrium. There is also evidence that the amount of scarring can predict ablation success rates. Recently, rapid ultra high density mapping equipment has become available and this has the capability of defining the electrical scar in the atrium in detail. The equipment used to do this is standard approved equipment for the procedure but its use for making scar maps has not been fully assessed.

In the mapping phase of the study therefore, the aim will be to collect high density scar maps in AF and normal rhythm to see how they compare. Maps will be collected in different ways to see if that changes their accuracy. The study will also assess if the values previously suggested as representing scar with lower density mapping systems are still appropriate where high density mapping equipment is used. The results from this study will help to improve the understanding of scar in the atrium and help demonstrate the most efficient way to collect scar information using this high density mapping equipment. In the future, clinicians may be able to use these very detailed scar maps to tailor and refine the way they ablate patients with AF, though the focus of the current study is just on collecting the scar information.

While identifying areas requiring ablation is important to an ablation procedure, the other important aspect is the efficacy of ablation. Until now, we have been reliant on assessing our inputs into an ablation (such as the level of contact and the power delivered) but have been limited in the assessment of the output of an ablation in terms of lesion characteristics. New ablation catheter technology is now available which can assess the localised impedance drop with ablation. This is likely a better surrogate for lesion parameters than what we have previously had available and merits further study. Based on such study, we may be able to define targets for ablation which would help to guide future ablations.

HD SAGA S:

Approval amendment March 2021 In addition to the above, using new catheter technology incorporating contact force into the assessment of ablation lesion efficacy.

HD SAGA H:

Approval amendment March 2021 Using new mapping catheter (HD Grid) and algorithms (HD Wave) to compare scar maps between AF and SR and pre-establish pulmonary vein isolation lines.

DETAILED DESCRIPTION:
HD SAGA:

The study would propose to use the Rhythmia Ultra High Density (UHD) mapping system (Boston Scientific) firstly to generate scar maps to determine if the results are comparable with previous work using lower density systems. Scar maps would be acquired in 3 groups of patients. The first group would be Redo-persistent AF ablation cases as these patients would have expected LA scar (iatrogenic and non-iatrogenic) from their previous ablation procedure. De novo persistent AF patients who would be expected to have non-iatrogenic scar. De novo paroxysmal AF patients who would be expected to have no or minimal scar. In redo AF patients, the validity of the scar maps would be further explored by undertaking re-isolation of veins based on discontinuities in the pulmonary vein isolation lines. If this is proven to be effective, it would demonstrate that the scar picked up by the system is genuine and may also suggest a more effective use of UHD systems for redo-pulmonary vein isolation (PVI).

In the ablation phase, we would be assessing the effect of ablation on the localised ablation characteristics of the tissue to assess how this is affected by ablation. From previous work, using conventional, wide area impedance measurements, there is a notable plateau in the impedance drop with ablation suggesting a point beyond which there is minimal efficacy gain from further ablation. One would expect this would be even more apparent with localised impedance.

Original Hypothesis - mapping phase An UHD mapping system can be utilised to generate automated, rapid, high density atrial scar maps in AF to guide a scar-based ablation strategy.

Original Hypothesis - ablation phase Localised Impedance will fall during ablation and this fall will plateau, suggesting a biophysical target for ablation

There is a small body of literature addressing contact mapping of atrial scar but this has mainly relied on lower density mapping approaches. UHD mapping systems offer the advantage of true high-density mapping with improved signal to noise ratios that one would predict will lead to the generation of more accurate maps. These advantages are also such that one would predict scar maps in AF would be more accurate. Extending the scar maps to incorporate the RA is also novel in this context and would give an insight into the degree to which AF is a bi-atrial fibrotic cardiomyopathy. As the use of UHD mapping is novel, it is important to establish how relevant criteria used in lower density, lower fidelity mapping systems are when the newer system is used, especially in defining scar.

No clinical studies have been published assessing localised impedance.

Protocol Fifteen patients listed for persistent AF ablation would be recruited including redo-ablation patients (aiming for 5 de novo and 10 redo patients). All these patients would be in AF at the time of the procedure. A further 5 patients with paroxysmal AF would also be recruited. Procedures would be performed on uninterrupted anticoagulation with a pre-procedural TOE as dictated by local guidelines. Moderate sedation or general anaesthetic procedures would be included. Intravenous heparin would be used to maintain the ACT at a therapeutic level throughout the study. All mapping would be undertaken using the Orion high density multipolar mapping catheter with the Rhythmia system. The ablation catheter used would be the IntellaNav MiFi Open Irrigated Temperature Ablation Catheter.

An RA scar map would be obtained using WCT as a reference. Double transseptal access would be obtained and the mapping and ablation catheters passed into the LA.

An LA scar map would be taken with the mapping catheter. For paroxysmal AF cases in sinus rhythm, this would be the only LA map taken. For patients in AF, maps would be taken in AF and then in sinus rhythm. In redo cases, the veins which the scar map suggests are likely to be reconnected would be noted (based on discontinuities in the wide area circumferential ablation (WACA) lines). The mapping catheter would then be used to confirm the presence of electrical reconnection of each vein. The patient would then be cardioverted if in AF and the mapping process repeated using a WCT reference. With all maps, the aim would be complete LA coverage. For the sinus rhythm maps, the LA will be divided into 5 sites: roof, posterior wall, inferior wall, septum, anterior wall bordering left atrial appendage. Within each of these sites, the pacing threshold will be assessed at 3 locations incorporating a spread of bipolar voltages.

Following the mapping phase, the case would then proceed as per the operator's standard methodology. The aim would be to collect at least 30 static study ablation points as discussed above. Vein re-isolation would be performed without any catheter measuring electrical activity in the vein, purely based on the scar map, targeting discontinuities in the WACA lines. Ablations would be static rather than drag ablations and at each point, the electrogram from the MiFi electrodes would be recorded at the start and end of ablation. Pacing would be performed during ablation and the impedance value at which pacing capture was lost would be noted. Following this ablation, the mapping catheter would be utilised to establish if the vein has been electrically disconnected based on the scar map.

At the end of the case, in sinus rhythm, scar maps of the RA would be taken. In sinus rhythm, pacing would be undertaken as for the LA at the following sites: anterior wall, posterior wall, septum and lateral wall.

The scar maps would be exported offline to allow quantitative analysis, as would the electrogram and impedance data. The analysis would be performed using the Matlab programming environment.

The scar analysis will exclude any portions of the LA distal to the WACA lines. The initial step will be to give a low voltage zone percentage. The next step will be to identify congruent low voltage zones and give advice regarding the ablation strategy for these - whether this involved delivering lines, for instance for a large posterior wall scar, and if the ablation needs to be extended to other inexcitable structures to prevent leaving a narrow conducting isthmus.

Study Follow up There would be no additional follow up for this study - the participants' follow up will follow the normal clinical practice at University Hospital Southampton.

HD SAGA S:

Protocol:

Twenty patients will be recruited for the HD-SAGAS cohort, all with persistent AF who will be in AF at the time of the procedure. These can be de novo or redo procedure patients.

Procedures would be performed on uninterrupted anticoagulation with a pre-procedural imaging as dictated by local guidelines. Moderate sedation or general anaesthetic procedures would be included. Intravenous heparin would be used to maintain the ACT at a therapeutic level throughout the study. All mapping would be undertaken using the Orion high density multipolar mapping catheter with the Rhythmia system. The ablation catheter used would be the Stablepoint catheter.

An LA scar map would be taken with the mapping catheter. The first map would be collected in AF. Following this, at 5 locations in the LA, aiming for a spread of voltages and locations, the contact force would be increased from 0-40g and the LI noted. The patient would then be cardioverted and a map taken in sinus rhythm with right atrial pacing. With all maps, the aim would be complete LA coverage. After cardioversion, at the same spots assessed in AF, the contact force would again be increased from 0-40g and the LI noted once more. Pacing thresholds would also be checked at these locations with a stable contact force of 10-20g to ensure good contact. The pacing phase could be after the ablation phase depending on rhythm stability.

Following the mapping phase, the case would then proceed as per the operator's standard methodology. The operator will be allowed to use whichever powers they wish to during ablation. Sites of acute reconnection would be noted.

At the end of the case, in sinus rhythm, pacing thresholds would be assessed in 5 areas in the LA, aiming for a spread of areas and voltages.

HD SAGA H:

The study would use the HD Grid catheter and Precision mapping system from Abbott. The HD Grid catheter has a unique arrangement of electrodes that allows for 3D electroanatomical maps to be generated between bipoles of different orientations. Following this a novel algorithm (HD Wave) provides the the point with largest amplitude. This abrogates the directional limitations of conventional bipolar mapping. Thus smaller more accurate areas of scar could be seen with the left atrium as has been generated in previous studies in the left ventricle.

Hypothesis The use of HD Wave mapping and the best duplicate algorithm will lead to more reliable voltage maps in AF - both throughout the LA body and in the PVI lines. The gold standard to compare with here will be the sinus rhythm maps.

Primary comparison:

Sinus rhythm HD wave versus AF HD wave map Scar volume PVI gaps

Secondary comparisons:

Scar volumes and PVI gaps Sinus rhythm HD wave versus conventional AF HD wave versus conventional

Protocol 20 patients listed for redo ablation of persistent AF, in AF at the time of procedure. All procedures would be performed using the precision mapping system.

The operator would collect a voltage map of the left atrium using the HD Grid catheter in AF. Following this, the patient would be cardioverted and another map collected with the same mapping catheter during CS proximal pacing.

The procedure would then proceed as per usual care. Subsequent to the procedure, the mapping functions would be applied to the data by Turbo mapping.

Sites of PV reconnection would be noted based on the ablations performed by the operator.

ELIGIBILITY:
Inclusion Criteria:

* trial Fibrillation, Scheduled for ablation on clinical grounds Able/willing to consent to procedure/research protocol No contraindication to clinical ablation

Exclusion Criteria:

* Unable/unwilling to consent Contraindication to clinical ablation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Scar Volume | Through study completion, an average of 1 year
  Quantification of scar volumes - presented as a proportion of the total atrial geometry volume
Impedance values with ablation | Through study completion, an average of 1 year
  Collection of localised and conventional impedance during ablation
Scar volume and pulmonary vein isolation line gaps | Through study completion, an average of 1 year
  Scar volume and pulmonary vein isolation line gaps between AF and SR

SECONDARY OUTCOMES:
Confirm Scar Thresholds | Through study completion, an average of 1 year
  Pacing threshold in mV will be assessed at different levels of atrial scar
Compare scar volumes in AF and sinus rhythm in the same patient | Through study completion, an average of 1 year
  Quantitative comparison - comparing the scar areas in cm2 between the two maps
Compare maps generated using internal unipolar reference and Wilson's Central Terminus | Through study completion, an average of 1 year
  Quantitative comparison - comparing the scar areas in cm2 between the two maps
Localised impedance fall during ablation | Through study completion, an average of 1 year
  Compare the LI fall versus time relationship to assess the nature of the relationship with the aim of generating a target for LI fall with ablation
Localised impedance fall versus electrogram attenuation | Through study completion, an average of 1 year
  Compare the LI impedance fall with ablation with electrogram attenuation (on microelectrodes) to further provide evidence for an LI target
Localised impedance fall versus pacing capture | Through study completion, an average of 1 year
  Compare the LI impedance fall with ablation with loss of acing capture during ablation to further provide evidence for an LI target
Compare localised with conventional impedance values during ablation | Through study completion, an average of 1 year
  Compare localised with conventional impedance values during ablation
Compare contact force measurements to local impedance | Through study completion, an average of 1 year
  Compare contact force (grams) measurements to local impedance (ohms) during ablation to establish if increasing levels of contact force result in greater local impedance drops
Compare left atrial scar area between omnipolar and bipolar mapping in atrial fibrillation | Through study completion, an average of 1 year
  Quantative comparison in cm2 of the level of atrial scar between 2 types of map in atrial fibrillation
Compare left atrial scar area between omnipolar and bipolar mapping in sinus rhythm | Through study completion, an average of 1 year
  Quantative comparison in cm2 of the level of atrial scar between 2 types of map in sinus rhythm
Compare left atrial scar area in omnipolar maps between sinus rhythm and atrial fibrillation | Through study completion, an average of 1 year
  Quantative comparison in cm2 of omnipolar maps between two heart rhythms
Compare left atrial scar areas in bipolar maps between sinus rhythm and atrial fibrillation | Through study completion, an average of 1 year
  Quantative comparison in cm2 of bipolar maps between two heart rhythms
Compare identification of pulmonary vein isolation gaps between omnipolar and bipolar maps | Through study completion, an average of 1 year
  Identifiying the presence of gaps within previously created pulmonary vein isolation lines between omnipolar and bipolar mapping
Compare identification of pulmonary vein isolation gaps between sinus rhythm and atrial fibrillation | Through study completion, an average of 1 year
  Identifiying the presence of gaps within previously created pulmonary vein isolation lines between different heart rhythms within the same patient

CONTACTS AND LOCATIONS:
Overall Officials: Waqas Ullah, PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD